CLINICAL TRIAL: NCT01222299
Title: Safety, Pharmacokinetics, and Efficacy of Bepotastine Besilate Nasal Product After Ragweed Pollen Exposure in an Environmental Chamber
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S00032
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 - Low Dose (Experimental): bepotastine besilate nasal product - low dose
  Interventions: Drug: bepotastine besilate nasal product - low dose
- Arm 2 - Medium Dose (Experimental): bepotastine besilate nasal product - medium dose
  Interventions: Drug: bepotastine besilate nasal product - medium dose
- Arm 3 - High Dose (Experimental): bepotastine besilate nasal product - high dose
  Interventions: Drug: bepotastine besilate nasal product - high dose
- Arm 4 - Placebo (Placebo Comparator): placebo comparator nasal product
  Interventions: Drug: placebo comparator nasal product

INTERVENTIONS:
Drug: bepotastine besilate nasal product - low dose — sterile nasal product
  Arms: Arm 1 - Low Dose
Drug: bepotastine besilate nasal product - medium dose — sterile nasal product
  Arms: Arm 2 - Medium Dose
Drug: bepotastine besilate nasal product - high dose — sterile nasal product
  Arms: Arm 3 - High Dose
Drug: placebo comparator nasal product — sterile nasal product
  Arms: Arm 4 - Placebo

SUMMARY:
The purpose of this study is to examine the safety and efficacy of bepotastine besilate nasal product in seasonal allergic rhinitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 to 65 years of age with a positive skin prick test with ragweed allergen

Exclusion Criteria:

* No active respiratory tract infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: placebo comparator nasal product
  placebo comparator nasal product: sterile nasal product twice daily
- Low Dose - 2%: bepotastine besilate nasal product - low dose
  bepotastine besilate nasal product - low dose: sterile nasal product twice daily
- Medium Dose - 4%: bepotastine besilate nasal product - medium dose
  bepotastine besilate nasal product - medium dose: sterile nasal product twice daily
- High Dose - 6%: bepotastine besilate nasal product - high dose
  bepotastine besilate nasal product - high dose: sterile nasal product twice daily
Period: Overall Study
Arm/Group | Placebo | Low Dose - 2% | Medium Dose - 4% | High Dose - 6%
Started | 21 | 23 | 22 | 23
Completed | 21 | 21 | 20 | 18
Not Completed | 0 | 2 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose - 2% | Medium Dose - 4% | High Dose - 6% | Total
Number analyzed (Participants) | 21 | 23 | 22 | 23 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (10.5) | 44.3 (9.5) | 42.1 (10.2) | 41.5 (10.7) | 42.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 12 | 11 | 46
  Male | 8 | 13 | 10 | 12 | 43

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (Pre-Dose) in Subject-rated Instantaneous TNSS
Description: Total nasal symptom scores (TNSS) was the summed scores for nasal pruritus [itching], rhinorrhea [runny nose], nasal congestion, and sneezing. Individual nasal symptoms were rated on a 4-point scale from 0-3 (0=Absent, 1=Mild, 2=Moderate, 3=Severe), with no half-unit assessments. TNSS was the sum score of 4 nasal symptoms with a maximum score for increased allergic response of 12 units. The minimum possible total score was 0.
Time Frame: Baseline, 20 days
Population: The per protocol population was based on participants who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose - 2% | Medium Dose - 4% | High Dose - 6%
Number analyzed (Participants) | 21 | 21 | 20 | 18
units on a scale
  Day 10 (after single dose) | -1.17 (1.88) | -0.69 (2.42) | -2.43 (2.73) | -1.65 (1.95)
  Day 20 (after twice daily dosing) | -1.63 (2.37) | -0.64 (2.93) | -2.52 (2.55) | -1.67 (2.22)

ADVERSE EVENTS:
Time Frame: 20 days
Arm/Group | Placebo | Low Dose - 2% | Medium Dose - 4% | High Dose - 6%
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/23 | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 7/21 | 9/23 | 9/22 | 11/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Low Dose - 2% (N=23) | Medium Dose - 4% (N=22) | High Dose - 6% (N=23)
Mild taste following instillation (General disorders) | 1 | 5 | 5 | 6
Headache (Nervous system disorders) | 4 | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.